CLINICAL TRIAL: NCT03422965
Title: Evaluation of Microvascular Changes in the Perifoveal Vascular Network Using Optical Coherence Tomography Angiography (OCT-A) in Type I Diabetes Mellitus
Brief Title: Perifoveal Vascular Network Assessed by OCT-Angiography in Type I Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Javier Zarranz-Ventura, MD, PhD, FEBO, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: OCTAMaratoTV3ICOF
Record Dates: First submitted 2018-01-24; First posted 2018-02-06 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Retinal Vascular; Retinal Disease; Retinal Ischemia; Retinal Ischaemia Due to Type 1 Diabetes Mellitus; Diabetes Mellitus; Diabetic Retinopathy; Diabetes Mellitus, Type 1; Vessels; Retina, Tortuous
Keywords: Retina; OCT; Optical Coherence Tomography; Optical Coherence Tomography Angiography; Systemic; Blood; Diabetes Mellitus; Diabetic Retinopathy
MeSH Terms: conditions — Retinal Diseases; Diabetes Mellitus; Diabetic Retinopathy; Diabetes Mellitus, Type 1 | interventions — Hematologic Tests; Urinalysis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 1 Diabetes Mellitus (Active Comparator): Cohort of Type 1 DM patients
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography; Diagnostic Test: Blood test; Diagnostic Test: Urine test
- Healthy controls (Sham Comparator): Cohort of Healthy controls
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography; Diagnostic Test: Blood test; Diagnostic Test: Urine test

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography Angiography — Optical Coherence Tomography Angiography images capture.
Diagnostic Test: Blood test — Blood test, systemic markers
Diagnostic Test: Urine test — Urine test, systemic markers

SUMMARY:
This study is directed to evaluate the role of Optical Coherence Tomography Angiography (OCT-A) in the evaluation of the perifoveal vascular network in type 1 diabetic patients, and to investigate the relationship between OCT-A-derived parameters and demographic and clinical factors, as metabolic control and duration of the disease.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is the leading cause of blindness in type 1 Diabetes Mellitus (DM) patients, as a consequence of impaired blood flow in the retina. Optical coherence tomography angiography (OCT-A) is a newly developed, non-invasive, retinal imaging technique that allows detection of perfused and non perfused areas of the retina without the injection of dye. This OCT-based method permits adequate delineation of the perifoveal vascular network, and allows objective identification of microvascular changes, such as capillary dilation or presence of microaneurisms. It is also capable to detect paramacular areas of capillary non perfusion and/or enlargement of the foveal avascular zone (FAZ), representing an excellent tool for assessment of diabetic retinopathy.

Given that all these features are commonly seen in diabetic patients, the relationship of these microvascular changes with systemic factors such as metabolic control or duration of the disease still need to be elucidated. Interestingly, further studies are required to investigate whether these changes reflect those occurring elsewhere in the body affected by diabetic microvascular disease, as the kidneys or the brain. If these relationships were demonstrated, early detection of these microvascular changes could lead to modifications in the pharmacological management of diabetic patients, as a way to reduce the risk of future complications in both the eye and other organs. The aim of this study is to evaluate the role of OCT-A in the evaluation of the perifoveal vascular network in type 1 diabetic patients, and to investigate the relationship between these OCT-A-derived parameters and demographic and clinical factors, as metabolic control and duration of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus
* Healthy controls

Exclusion Criteria:

* Ocular pathologies other than diabetic retinopathy (i.e. age-related macular degeneration, retinal vein occlusions, uveitis, glaucoma, etc.)
* Axial length: <-6.00 to >+3.00 diopters
* Media Opacities
* Unability to capture OCT images

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2021-03-08 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Perifoveal vessel density | 24 months
  OCTA images will be processed to obtain vascular density measurements in this area (mm-1)

SECONDARY OUTCOMES:
Parafoveal vessel density | 24 months
  OCTA images will be processed to obtain vascular density measurements in this area (mm-1)
Total Avascular Area | 24 months
  OCTA images will be processed to obtain total avascular area measurements (mm2)
Foveal Avascular Zone | 24 months
  OCTA images will be processed to obtain foveal avascular zone area measurements (mm2)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Zarranz-Ventura, MD PhD FEBO, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Institut Clinic de Oftalmologia (ICOF), Hospital Clínic de Barcelona, Barcelona
  - Diabetes Unit, Institut Clinic de Malalties Digestives i Métaboliques (ICMDM), Hospital Clínic de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Song SJ, Wong TY. Current concepts in diabetic retinopathy. Diabetes Metab J. 2014 Dec;38(6):416-25. doi: 10.4093/dmj.2014.38.6.416. PMID 25541604
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. II. Prevalence and risk of diabetic retinopathy when age at diagnosis is less than 30 years. Arch Ophthalmol. 1984 Apr;102(4):520-6. doi: 10.1001/archopht.1984.01040030398010. PMID 6367724
- [Background] Shah CA. Diabetic retinopathy: A comprehensive review. Indian J Med Sci. 2008 Dec;62(12):500-19. PMID 19265246
- [Background] Roser P, Kalscheuer H, Groener JB, Lehnhoff D, Klein R, Auffarth GU, Nawroth PP, Schuett F, Rudofsky G. Diabetic Retinopathy Screening Ratio Is Improved When Using a Digital, Nonmydriatic Fundus Camera Onsite in a Diabetes Outpatient Clinic. J Diabetes Res. 2016;2016:4101890. doi: 10.1155/2016/4101890. Epub 2016 Jan 21. PMID 26904690
- [Background] Looker HC, Nyangoma SO, Cromie DT, Olson JA, Leese GP, Philip S, Black MW, Doig J, Lee N, Briggs A, Hothersall EJ, Morris AD, Lindsay RS, McKnight JA, Pearson DW, Sattar NA, Wild SH, McKeigue P, Colhoun HM; Scottish Diabetes Research Network (SDRN) Epidemiology Group and the Scottish Diabetic Retinopathy Collaborative. Predicted impact of extending the screening interval for diabetic retinopathy: the Scottish Diabetic Retinopathy Screening programme. Diabetologia. 2013 Aug;56(8):1716-25. doi: 10.1007/s00125-013-2928-7. Epub 2013 May 21. PMID 23689796
- [Background] Zimmer-Galler IE, Kimura AE, Gupta S. Diabetic retinopathy screening and the use of telemedicine. Curr Opin Ophthalmol. 2015 May;26(3):167-72. doi: 10.1097/ICU.0000000000000142. PMID 25759962
- [Background] Gass JD. A fluorescein angiographic study of macular dysfunction secondary to retinal vascular disease. IV. Diabetic retinal angiopathy. Arch Ophthalmol. 1968 Nov;80(5):583-91. doi: 10.1001/archopht.1968.00980050585004. No abstract available. PMID 5684307
- [Background] Fioretto P, Mauer M, Brocco E, Velussi M, Frigato F, Muollo B, Sambataro M, Abaterusso C, Baggio B, Crepaldi G, Nosadini R. Patterns of renal injury in NIDDM patients with microalbuminuria. Diabetologia. 1996 Dec;39(12):1569-76. doi: 10.1007/s001250050616. PMID 8960844
- [Background] Kwiterovich KA, Maguire MG, Murphy RP, Schachat AP, Bressler NM, Bressler SB, Fine SL. Frequency of adverse systemic reactions after fluorescein angiography. Results of a prospective study. Ophthalmology. 1991 Jul;98(7):1139-42. doi: 10.1016/s0161-6420(91)32165-1. PMID 1891225
- [Background] Yeung L, Lima VC, Garcia P, Landa G, Rosen RB. Correlation between spectral domain optical coherence tomography findings and fluorescein angiography patterns in diabetic macular edema. Ophthalmology. 2009 Jun;116(6):1158-67. doi: 10.1016/j.ophtha.2008.12.063. Epub 2009 Apr 23. PMID 19395034
- [Background] Jia Y, Tan O, Tokayer J, Potsaid B, Wang Y, Liu JJ, Kraus MF, Subhash H, Fujimoto JG, Hornegger J, Huang D. Split-spectrum amplitude-decorrelation angiography with optical coherence tomography. Opt Express. 2012 Feb 13;20(4):4710-25. doi: 10.1364/OE.20.004710. PMID 22418228
- [Background] Jia Y, Bailey ST, Hwang TS, McClintic SM, Gao SS, Pennesi ME, Flaxel CJ, Lauer AK, Wilson DJ, Hornegger J, Fujimoto JG, Huang D. Quantitative optical coherence tomography angiography of vascular abnormalities in the living human eye. Proc Natl Acad Sci U S A. 2015 May 5;112(18):E2395-402. doi: 10.1073/pnas.1500185112. Epub 2015 Apr 20. PMID 25897021
- [Background] Ishibazawa A, Nagaoka T, Takahashi A, Omae T, Tani T, Sogawa K, Yokota H, Yoshida A. Optical Coherence Tomography Angiography in Diabetic Retinopathy: A Prospective Pilot Study. Am J Ophthalmol. 2015 Jul;160(1):35-44.e1. doi: 10.1016/j.ajo.2015.04.021. Epub 2015 Apr 18. PMID 25896459
- [Background] de Carlo TE, Chin AT, Bonini Filho MA, Adhi M, Branchini L, Salz DA, Baumal CR, Crawford C, Reichel E, Witkin AJ, Duker JS, Waheed NK. DETECTION OF MICROVASCULAR CHANGES IN EYES OF PATIENTS WITH DIABETES BUT NOT CLINICAL DIABETIC RETINOPATHY USING OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY. Retina. 2015 Nov;35(11):2364-70. doi: 10.1097/IAE.0000000000000882. PMID 26469537
- [Background] Takase N, Nozaki M, Kato A, Ozeki H, Yoshida M, Ogura Y. ENLARGEMENT OF FOVEAL AVASCULAR ZONE IN DIABETIC EYES EVALUATED BY EN FACE OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY. Retina. 2015 Nov;35(11):2377-83. doi: 10.1097/IAE.0000000000000849. PMID 26457396
- [Background] Hwang TS, Gao SS, Liu L, Lauer AK, Bailey ST, Flaxel CJ, Wilson DJ, Huang D, Jia Y. Automated Quantification of Capillary Nonperfusion Using Optical Coherence Tomography Angiography in Diabetic Retinopathy. JAMA Ophthalmol. 2016 Apr;134(4):367-73. doi: 10.1001/jamaophthalmol.2015.5658. PMID 26795548
- [Derived] Rosines-Fonoll J, Martin-Pinardel R, Marias-Perez S, Suarez-Valero X, Feu-Basilio S, Marin-Martinez S, Bernal-Morales C, Castro-Dominguez R, Mendez-Mourelle A, Oliva C, Vila I, Hernandez T, Vinagre I, Mateu-Salat M, Ortega E, Gimenez M, Zarranz-Ventura J. Optical Coherence Tomography Angiography in Type 1 Diabetes Mellitus. Report 5: Cardiovascular Risk. Biomedicines. 2026 Jan 11;14(1):153. doi: 10.3390/biomedicines14010153. PMID 41595687
- [Derived] Toha-Dalmau A, Rosines-Fonoll J, Romero E, Mazzanti F, Martin-Pinardel R, Marias-Perez S, Bernal-Morales C, Castro-Dominguez R, Mendez A, Ortega E, Vinagre I, Gimenez M, Vellido A, Zarranz-Ventura J. Machine Learning Prediction of Cardiovascular Risk in Type 1 Diabetes Mellitus Using Radiomic Features from Multimodal Retinal Images. Ophthalmol Sci. 2025 Jul 4;5(6):100874. doi: 10.1016/j.xops.2025.100874. eCollection 2025 Nov-Dec. PMID 40893617
- [Derived] Sala-Vila A, Vinagre I, Cofan M, Lazaro I, Ale-Chilet A, Barraso M, Hernandez T, Harris WS, Zarranz-Ventura J, Ortega E. Blood omega-3 biomarkers, diabetic retinopathy and retinal vessel status in patients with type 1 diabetes. Eye (Lond). 2025 Jun;39(8):1526-1531. doi: 10.1038/s41433-025-03705-5. Epub 2025 Feb 18. PMID 39966603
- [Derived] Carrera-Escale L, Benali A, Rathert AC, Martin-Pinardel R, Bernal-Morales C, Ale-Chilet A, Barraso M, Marin-Martinez S, Feu-Basilio S, Rosines-Fonoll J, Hernandez T, Vila I, Castro-Dominguez R, Oliva C, Vinagre I, Ortega E, Gimenez M, Vellido A, Romero E, Zarranz-Ventura J. Radiomics-Based Assessment of OCT Angiography Images for Diabetic Retinopathy Diagnosis. Ophthalmol Sci. 2022 Nov 21;3(2):100259. doi: 10.1016/j.xops.2022.100259. eCollection 2023 Jun. PMID 36578904
- [Derived] Bernal-Morales C, Ale-Chilet A, Martin-Pinardel R, Barraso M, Hernandez T, Oliva C, Vinagre I, Ortega E, Figueras-Roca M, Sala-Puigdollers A, Gimenez M, Esmatjes E, Adan A, Zarranz-Ventura J. Optical Coherence Tomography Angiography in Type 1 Diabetes Mellitus. Report 4: Glycated Haemoglobin. Diagnostics (Basel). 2021 Aug 25;11(9):1537. doi: 10.3390/diagnostics11091537. PMID 34573883
- [Derived] Barraso M, Ale-Chilet A, Hernandez T, Oliva C, Vinagre I, Ortega E, Figueras-Roca M, Sala-Puigdollers A, Esquinas C, Esmatjes E, Adan A, Zarranz-Ventura J. Optical Coherence Tomography Angiography in Type 1 Diabetes Mellitus. Report 1: Diabetic Retinopathy. Transl Vis Sci Technol. 2020 Sep 30;9(10):34. doi: 10.1167/tvst.9.10.34. eCollection 2020 Sep. PMID 33062397
- [Derived] Zarranz-Ventura J, Barraso M, Ale-Chilet A, Hernandez T, Oliva C, Gascon J, Sala-Puigdollers A, Figueras-Roca M, Vinagre I, Ortega E, Esmatjes E, Adan A. Evaluation of microvascular changes in the perifoveal vascular network using optical coherence tomography angiography (OCTA) in type I diabetes mellitus: a large scale prospective trial. BMC Med Imaging. 2019 Nov 21;19(1):91. doi: 10.1186/s12880-019-0391-8. PMID 31752726